CLINICAL TRIAL: NCT01523925
Title: Combined Behavioral Approaches With Functional Electrical Therapy in Stroke Rehabilitation: Effects on Motor Control, Motor Impairment, Daily Function and Community Reintegration
Brief Title: Combined Behavioral Approaches With Functional Electrical Therapy in Stroke Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NSC 99-2314-B-182-014-MY3; 98-3827B (Other: Chang Gung Memorial Hospital)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2014-09

CONDITIONS: Cerebrovascular Accident
Keywords: Functional electrical therapy; Bilateral arm training; Constraint induced therapy; Stroke rehabilitation; Clinical evaluation; Kinematic analysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Combined dCIT with FET (Experimental): Combined distributed constraint induced therapy with functional electrical therapy
  Interventions: Behavioral: dCIT; Behavioral: Functional electrical stimulation
- Combined BAT with FET (Experimental): Combined bilateral arm treatment with functional electrical therapy
  Interventions: Behavioral: BAT; Behavioral: Functional electrical stimulation
- Control intervention group (Active Comparator): Control intervention
  Interventions: Behavioral: Control intervention group
- dCIT (Experimental): distributed constraint induced therapy
  Interventions: Behavioral: dCIT
- BAT (Experimental): bilateral arm treatment
  Interventions: Behavioral: BAT

INTERVENTIONS:
Behavioral: dCIT — This dCIT group focuses on restriction on movement of the unaffected hand by placement of the hand in a mitt for 6 hours/day and intensive training of the affected upper extremity in functional tasks 1.5 hours/weekday, for 4 weeks. The level of challenge will be adapted based on patient ability and improvement during training. Patients will be encouraged to initiate the designed therapeutic functional activities.
  Other Names: distributed constraint induced therapy
  Arms: Combined dCIT with FET; dCIT
Behavioral: BAT — The BAT group concentrates on the simultaneous movements of both the affected and unaffected upper extremity on robot for 1.5 hours/day, 5 days/week for 4 weeks.
  Other Names: bilateral arm training
  Arms: BAT; Combined BAT with FET
Behavioral: Control intervention group — The conventional intervention group is designed to control for the duration and intensity of patient-therapist interactions and therapeutic activities (1.5 hours/day, 5 days/week, for 4 weeks). Therapy in the control intervention group will involve training for coordination, balance, and movements of the affected upper extremity, as well as compensatory practice on functional tasks with the unaffected upper extremity or both upper extremities.
  Other Names: Control intervention
  Arms: Control intervention group
Behavioral: Functional electrical stimulation
  Other Names: FES
  Arms: Combined BAT with FET; Combined dCIT with FET

SUMMARY:
This project attempts to perform a randomized controlled trial to verify the efficacy and motor control mechanism of the proposed combined functional electrical therapy with distributed constraint-induced therapy or with robot-assisted Bilateral training.

DETAILED DESCRIPTION:
Two theory-based, task-oriented approaches are distributed CIT (dCIT) and robot-assisted Bilateral training(BAT). CIT/dCIT involves massed practice of the affected arm and restraint of the unaffected arm. BAT involves repetitive practice of symmetrical bilateral movements on robot. Both are evident to improve motor performance, motor control or daily function in high functioning patients. These dCIT and BAT have their own limitations for motor-deficit rehabilitation after stroke, i.e. only appropriate for high-functioning or mildly motor impaired patients. Functional electrical therapy, an innovative technology, is proposed as an adjunct to these behavioral approaches to assist in movement execution. Functional electrical therapy is used to increase the electric activity of muscles for movement and the active range of motion in low functioning patients. Combining functional electrical therapy into CIT or BAT may extend the utility of these two behavioral approaches beyond patients with mild motor deficits and could expedite the progress of motor recovery. This project attempts to perform a randomized controlled trial to verify the efficacy and motor control mechanism of the proposed combined functional electrical therapy with dCIT or with BAT.

ELIGIBILITY:
Inclusion Criteria:

* The onset duration more than 6 months
* An initial upper extremity subsection of the Fugl-Meyer Assessment score of 33 to 52 indicating moderate or moderate-to-mild movement impairment
* No serious cognitive deficits (a score of more than 24 on the Mini Mental State Exam)
* The availability of caregiver for assistance during the 6-hour restraint time of unaffected extremity per day
* No balance problems sufficient to compromise safety when wearing the project's constraint device with the assistance of the caregiver
* Considerable nonuse of the affected upper extremity (an AOU score < 2.5 of Motor Activity Log)

Exclusion Criteria:

* Exhibit physician determined major medical problems or poor physical conditions that would interfere with participation
* Excessive pain in any joint that might limit participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Movement time (MT) | Baseline and change from baseline in MT at 4 weeks
  The movement time is collected by a 7-camera motion analysis system (VICON MX 3-D, Oxford Metrics Inc., Oxford, UK) from unilateral and bilateral reaching tasks of pressing the desk bell. MT is the interval between movement onset and offset.
Total displacement (TD) | Baseline and change from baseline in TD at 4 weeks
  The movement time is collected by a 7-camera motion analysis system (VICON MX 3-D, Oxford Metrics Inc., Oxford, UK) from unilateral and bilateral reaching tasks of pressing the desk bell. TD refers to the path of a hand in three-dimensional space and is a measure of trajectory smoothness.
Percentage of peak velocity (PPV) | Baseline and change from baseline in PPV at 4 weeks
  The movement time is collected by a 7-camera motion analysis system (VICON MX 3-D, Oxford Metrics Inc., Oxford, UK) from unilateral and bilateral reaching tasks of pressing the desk bell. The PPV reflects the duration of the acceleration phase relative to the deceleration phase and indicates the type of movement strategy selected for a motor action.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline, change from baseline in FMA at 2 weeks, and change from baseline in FMA at 4 weeks
  The UE subscale of the FMA (max. score 66) uses a 3-point ordinal scale to assess motor impairment.
Medical Research Council scale (MRC) | Baseline, change from baseline in MRC at 2 weeks, and change from baseline in MRC at 4 weeks
  The MRC scale examines the muscle strength of the affected arm and is reliable measurement with score ranged from 0 (no contraction) to 5 (normal power).
Modified Ashworth Scale (MAS) | Baseline, change from baseline in MAS at 2 weeks, and change from baseline in MAS at 4 weeks
  The MAS scale is an ordinal scale (0-5 points) assessing spasticity of skeletal muscle in UE. A higher score indicating more spasticity.
MYOTON-3 | Baseline, change from baseline in MYOTON-3 at two weeks, and change from baseline in MYOTON-3 at 4 weeks
  Assessment of the functional state of skeletal muscle was carried out using myometric measurements with the MYOTON-3 device.
Motor Activity Log (MAL) | Baseline, change of MAL at 2 weeks, and change of MAL at 4 weeks
  The MAL is a semi-structured interview of patients to assess the amount of use (AOU) and quality of movement (QOM) of the affected upper extremity in 30 important daily activities using a 6-point ordinal scale. Higher scores indicate better performance.
ABILHAND Questionnaire | Baseline, change of ABILHAND Questionnaire at 2 weeks, and change of ABILHAND Questionnaire at 4 weeks
  ABILHAND questionnaire is an inventory of 56 manual activities that uses a 3-point ordinal scale to measure subjectively perceived difficulty in performing everyday bimanual activity.
Reintegration of Normal Living Index (RNL) | Baseline, change of RNL at 2 weeks, and change of RNL at 4 weeks
  The RNL is used to measure the satisfaction with community reintegration. It scores on a 4-point ordinal scale, with higher scores indicating a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan